CLINICAL TRIAL: NCT06585332
Title: Hand Grip Strength As a Screening Tool for Respiratory Dysfunction in Huntington's Disease
Brief Title: Handgrip and Respiratory Dysfunction in HD Patients.
Status: Completed | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Romana Konvalinková, physiotherapist of the rehabilitation section in General University Hospital Prague, General University Hospital, Prague
Other Study IDs: HGS IPD Resp HD
Record Dates: First submitted 2024-08-28; First posted 2024-09-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-09

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Respiratory dysfunction; Peak cough flow; Handgrip strength; Screening tool
MeSH Terms: conditions — Huntington Disease; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons with HD: One group - adult patients with genetically confirmed Huntington disease.
  Interventions: Other: Assessment of respiratory paramenters (Maximal inspiratory pressure, maximal expiratory pressure, and voluntary peak cough flow))

INTERVENTIONS:
Other: Assessment of respiratory paramenters (Maximal inspiratory pressure, maximal expiratory pressure, and voluntary peak cough flow)) — The voluntary peak cough flow is measured using a pneumotachograph (BTL cardiopoint Spiro, BTL industries), which meets the recommendations of the American Thoracic Society and the European Respiratory Society for range and accuracy in forced expiratory maneuvers.
  Maximal expiratory and inspiratory pressures assessments were performed using a flanged rubber mouthpiece connected to a pressure manometer (Micro RPM, Vyaire Medical). Assessments are conducted according to the statements on respiratory muscle testing of the American Thoracic Society and the European Respiratory Society.
  Hand grip strength Grip strength is measured using DHD-1 digital hand dynamometer (SAEHAN®,Seahan Corporation), assessment follows recommendation of The American Society of Hand Therapists.
  Other Names: Assessment of hand grip strength; Questionnaire: Index of pulmonary dysfunction

SUMMARY:
Hereditary neurodegenerative diagnosis of Huntington's disease (HD) is associated with a progressive deterioration of the respiratory system function . This fact contributes strongly to the increased risk of aspiration pneumonia as a primary cause of death in people with HD. But regularly objective monitoring of the airway system condition is in common clinical practice almost impossible for high time requirements and the need for specialized expensive devices . This drives the need for a simpler and more cost-effective screening tool. In recent years published studies, working with all ages and genders, show correlation between hand grip strength (HGS) and respiratory parameters. As a second simple screening tool, we chose a short questionnaire called the Index of pulmonary dysfunction.

DETAILED DESCRIPTION:
Goal: To identify a simple method for screening respiratory muscle and cough weakness in Huntington's Disease (HD) patients, suitable for clinical practice.

Hypothesis 1: Maximal inspiratory pressure, maximal expiratory pressure, and voluntary peak cough flow will be significantly correlated with maximal hand grip strength in HD patients.

Hypothesis 2: Maximal inspiratory pressure, maximal expiratory pressure, and voluntary peak cough flow will be significantly correlated with the Index of pulmonary dysfunction in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmed diagnosis of Huntington's disease

Exclusion Criteria:

* diagnosis of other concomitant neurological diseases;
* a history of cardiovascular or lung disease;
* respiratory symptoms such as cough, phlegm, wheezing, or dyspnea at the time of assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with confirmed diagnosis of Huntington's disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Maximal Hand grip strength | Up to 35 weeks (once on a single screening visit)
  Unit of Measure: kg Assessment followed recommendation of The American Society of Hand Therapists. HSG is measured using DHD-1 digital hand dynamometer (SAEHAN®,Seahan Corporation).
Voluntary peak cough flow | Up to 35 weeks (once on a single screening visit)
  Unit of measure: l/min Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Maximal expiratory pressure, Maximal inspiratory pressure | Up to 35 weeks (once on a single screening visit)
  Unite of measure: cmH2O Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

SECONDARY OUTCOMES:
Index of Pulmonary dysfunction | Up to 35 weeks (once on a single screening visit)
  Questionnaire of four questions. Scale range: 0-11 points A higher score indicates a worse pulmonary condition.

CONTACTS AND LOCATIONS:
Overall Officials: Romana Konvalinkova, MS, Principal Investigator — General University Hospital
Locations (1):
- General University Hospital, Prague, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones U, Busse M, Enright S, Rosser AE. Respiratory decline is integral to disease progression in Huntington's disease. Eur Respir J. 2016 Aug;48(2):585-8. doi: 10.1183/13993003.02215-2015. Epub 2016 Jun 23. PMID 27338194
- [Background] Reyes A, Cruickshank T, Ziman M, Nosaka K. Pulmonary function in patients with Huntington's disease. BMC Pulm Med. 2014 May 26;14:89. doi: 10.1186/1471-2466-14-89. PMID 24886346
- [Background] Schumann-Werner B, Dogan I, Mirzazade S, Mall B, Overbeck R, Honrath P, Schulz JB, Reetz K, Werner CJ. Clinical predictors and neural correlates for compromised swallowing safety in Huntington disease. Eur J Neurol. 2021 Sep;28(9):2855-2862. doi: 10.1111/ene.14953. Epub 2021 Jun 24. PMID 34077591
- [Background] Jakusova J, Brozmanova M. Methods of Cough Assessment and Objectivization. Physiol Res. 2023 Dec 31;72(6):687-700. doi: 10.33549/physiolres.935062. PMID 38215057
- [Background] Ohara DG, Pegorari MS, Oliveira Dos Santos NL, de Fatima Ribeiro Silva C, Monteiro RL, Matos AP, Jamami M. Respiratory Muscle Strength as a Discriminator of Sarcopenia in Community-Dwelling Elderly: A Cross-Sectional Study. J Nutr Health Aging. 2018;22(8):952-958. doi: 10.1007/s12603-018-1079-4. PMID 30272099
- [Background] Efstathiou ID, Mavrou IP, Grigoriadis KE. Correlation Between Maximum Inspiratory Pressure and Hand-Grip Force in Healthy Young and Middle-Age Individuals. Respir Care. 2016 Jul;61(7):925-9. doi: 10.4187/respcare.04319. Epub 2016 Apr 19. PMID 27094394
- [Background] Shin HI, Kim DK, Seo KM, Kang SH, Lee SY, Son S. Relation Between Respiratory Muscle Strength and Skeletal Muscle Mass and Hand Grip Strength in the Healthy Elderly. Ann Rehabil Med. 2017 Aug;41(4):686-692. doi: 10.5535/arm.2017.41.4.686. Epub 2017 Aug 31. PMID 28971054
- [Background] Bahat G, Tufan A, Ozkaya H, Tufan F, Akpinar TS, Akin S, Bahat Z, Kaya Z, Kiyan E, Erten N, Karan MA. Relation between hand grip strength, respiratory muscle strength and spirometric measures in male nursing home residents. Aging Male. 2014 Sep;17(3):136-40. doi: 10.3109/13685538.2014.936001. Epub 2014 Jul 4. PMID 24993454
- [Background] Enright PL, Kronmal RA, Manolio TA, Schenker MB, Hyatt RE. Respiratory muscle strength in the elderly. Correlates and reference values. Cardiovascular Health Study Research Group. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):430-8. doi: 10.1164/ajrccm.149.2.8306041.
- [Background] Srp M, Bartosova T, Klempir J, Lagnerova R, Gal O, Listvanova T, Jech R, Ruzicka E, Hoskovcova M. Expiratory Muscle Strength Training in Multiple System Atrophy: A Pilot Study. Mov Disord Clin Pract. 2023 May 19;10(7):1060-1065. doi: 10.1002/mdc3.13765. eCollection 2023 Jul. PMID 37476315
- [Background] Smeltzer SC, Lavietes MH, Troiano R, Cook SD. Testing of an Index of Pulmonary Dysfunction in Multiple Sclerosis. Nurs Res. 1989 Nov-Dec;38(6):370-4. PMID 2587294
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Derived] Konvalinkova R, Srp M, Doleckova K, Capek V, Gal O, Hoskovcova M, Klempir J. Handgrip strength and the Index of pulmonary dysfunction: Practical screening tools for cough dysfunction in huntington's disease. J Huntingtons Dis. 2026 Feb;15(1):148-155. doi: 10.1177/18796397251385607. Epub 2025 Oct 14. PMID 41332279